| Regular home use of dual-light photodynamic therapy as an adjunct | to |
|-------------------------------------------------------------------|----|
| non-surgical periodontal treatment in smokers | |

10.16.22

## Clinical investigation plan (CIP)

| Regular home use of dual-light photodynamic therapy as adjunct to non-surgical periodontal treatment in smokers | Pages | |
|---|---|---|
| Study code: Thss1 | Version<br>FINAL | Date |

| Revision | Change details and rationale | Author/Effective | Accepted |
|----------|------------------------------|-------------------|----------|
| No. | | date | |
| 1. | First version | Tommi Pätilä | |
| 2. | Second version | Dimitra Sakellari | |
| | | Aikaterini- | |
| | | Elisavet Doufexi | |
| | | Chrysoula Vakaki | |

**Principal investigator:** Dimitra Sakellari, Professor

Department of Preventive Dentistry, Periodontology and Implant

Biology,(AUTh) · Aristotle University of Thessaloniki Central Office, A' basement Zip code 54124, Thessaloniki

Tel. +

mailto:dimisak@gmail.com

**Coordinating investigator:** Timo Sorsa, Professor

University of Helsinki

Department of Oral and Maxillofacial Diseases

Biomedicum 1 Helsinki, Haartmaninkatu 8 00290 Helsinki,

Finland, Tel. +358 504151327/ +358 294127294

email: timo.sorsa@helsinki.fi

**Investigators:** This project will serve as the M.Sc thesis of the 2<sup>nd</sup> year

postgraduate student, Chrysoula Vakaki, at the Department of Preventive Dentistry, Periodontology and Implant Biology Chrysoula Vakaki, Periodontist, <a href="mailto:vakakichri@gmail.com">vakakichri@gmail.com</a>

Aikaterini-Elisavet Doufexi, Assistant

Professor, vdoufexi@yahoo.com

Ismo Räisänen, PhD, <u>ismo.raisanen@helsinki.fi</u>
Tommi Pätilä, MD, PhD <u>tommi.patila@gmail.com</u>

Investigational site: Department of Preventive Dentistry, Periodontology and Implant

Biology, (AUTh) · Aristotle University of Thessaloniki Central Office, A' basement Zip code 54124, Thessaloniki

Other institutions: University of Helsinki

Department of Oral and Maxillofacial Diseases Biomedicum 1 Helsinki, Haartmaninkatu 8,

00290 Helsinki, Finland

## Overall synopsis of the clinical investigation

**Study title:** Regular home use of dual-light photodynamic therapy as an adjunct to non-surgical periodontal treatment in smokers

**Type:** Investigator initiated study

**Study Center**: Department of Preventive Dentistry, Periodontology and Implant Biology, (AUTh) · Aristotle University of Thessaloniki

Name of the Investigational Medical Device (IMD): 1) Lumoral treatment device 2) Lumorinse mouth rinse

Manufacturer of the Investigational Device: Koite Health Oy, Kutojantie 2 C, 02630 Espoo

Study code: Thss1

**Investigators and the study center:** Principal Investigator: Dimitra Sakellari; Coordinating Investigator: Timo Sorsa; Investigators: Chrysoula Vakaki, Aikaterini- Elisavet Doufexi, Ismo Räisänen, Tommi Pätilä

Study initiation and ending date: 01.09.2022 to 01.09.24

**Objectives:** To investigate the impact of regular home use of Lumoral device as an adjunct treatment compared to non-surgical periodontitis treatment alone on biofilm removal and host response in Stage III and Grade C smoking periodontitis patients at 3 months.

Methodology: Randomized study; randomization method: www.randomizer.org

**Sample size:** 60 subjects, 30 subjects in the study group, and 30 in the control group. The subjects have a referral to visit a specialist dentist/ periodontist

Main criteria for inclusion: Periodontal disease Stage III and Grade C with at least 6 sites with probing depth (PD) and clinical attachment loss (CAL)  $\geq$ 5 mm and bleeding on probing (BOP)  $\geq$ 15 teeth; aged  $\geq$ 35; smokers smoking $\geq$ 10 cigarettes per day, at least 18 years old, presence of  $\geq$ 20 teeth, agreement to participate in the study and a written consent form signed.

Main criteria for exclusion: Presence of any physical limitation or restriction that might restrict Lumoral use, need for prophylactic antimicrobial coverage; scaling and root planing performed during the previous 6 months; non-smoking status or smoking less than 10 cigarettes per day; antimicrobial therapy in the previous 6 months; immune modifying conditions/ diseases (e.g., diabetes mellitus, rheumatoid arthritis, and osteoporosis); long-term use of medication that could interfere with periodontal response (e.g., bisphosphonates); pregnancy or lactation.

Estimated duration of the data gathering in the clinical investigation: 6 months

Assessments:

Primary outcome: Difference in the number of reduced deep pockets (i.e. PD≤ 4mm, no BOP) between the test and the control group.

Secondary outcome: PD, CAL, BOP, Turetsky Modified Quigley-Hein Plaque Index (TMQHPI), levels of MMP-8, and Oral Health Quality of Life (OHQL). Need for optional SRP

Statistical methods: Wilcoxon test, Mann-Whitney U-test, Fisher's test, Pearson's correlation test

## Study flowchart/ Schedule of visits and study procedures



| Visit #/code | 1 | 2 | 3 | 4 | 5 | Х |
|---|---|---|---|---|---|---|
| | | 6 | 2 16 11 | 40 | 2 ( !! | |
| Reason for visit | Screening/<br>Baseline/ | Start of the intervention | 2-week follow-<br>up/ SRP in 2<br>sessions in 2<br>weeks | 10<br>-week<br>follow-up | 3 month follow-<br>up | Termination |
| Inclusion/ exclusion criteria | х | | | | | |
| Informed consent | x | | | | | |
| Subject ID | х | | | | | |
| Subject demography | х | | | | | |
| Medications (changes*) | х | | | | x* | |
| Oral and general disease history (changes*) | Х | | | | х* | |
| Assessments | | | | | | |
| aMMP-8 sampling | | x | х | x | х | |
| (oral rinse) | | | | | | |
| Potential Microbial | | х | | × | х | |
| sampling<br>(periodontal<br>pocket) | | | | | | |
| Full mouth X-rays | х | | | | | |
| BOP% | | х | | Х | х | |
| TMQHPI % | | х | х | х | х | |
| PPD | | х | | х | х | |
| CAL | | х | | Х | х | |
| Oral hygiene instructions | | х | х | х | х | |
| Lumoral instructions (only study group) | | х | х | Х | х | |
| Lumoral diary for use (only study group) | | х | х | Х | х | |
| Reason for termination | | | | | | Х |
| AE/ADE/SAE/<br>SADE/DD | | | Х | х | Х | Х |

## **Power Calculation**

Previous results showed statistically significant changes in plaque development in 15 patients in a randomized, split-mouth study (Nikinmaa et al. 2021a). In this clinical study plan, more effective antibacterial therapy shall be used. According to our published laboratory analysis, the dual-light antibacterial treatment would be at least a 3-log scale more potent than the treatment used in the split-mouth protocol (Nikinmaa 2021). In another pilot study in peri-implant patients using this more effective treatment, a significant change in plaque was already observed in the data of seven patients during four weeks of Lumoral treatment (Lähteenmäki et al., 2022).

Based on this limited but promising available data, a power calculation (SAS 9.4, Cary, NC, USA) was performed and levels for 5% alpha error and 20% TYPE II error (80% power) were determined. It was

concluded that the sample size of 25 patients in each study arm was sufficient to allow statistical calculations. 30 + 30 patients were assigned to cover possible dropouts.



Total time: 24 weeks from time 0